CLINICAL TRIAL: NCT02233777
Title: Bioequivalence Study of 150 mg Pregabalin Capsules Produced by PT Dexa Medica in Comparison With the Comparator Product (Lyrica® Capsule 150 mg, Pfizer Manufacturing Deutschland GmbH, Germany)
Brief Title: Bioequivalence Study of Two Formulations of Pregabalin Capsules 150 mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BE.293/EQL/2013
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Pregabalin; Bioequivalence; Bioavailability; Pharmacokinetic; Antiepileptic
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin capsules 150 mg of Dexa Medica (Experimental): Each capsule contains 150 mg pregabalin.
  Interventions: Drug: Pregabalin capsules 150 mg of Dexa Medica
- Pregabalin capsules 150 mg of Pfizer Manufacturing Deutschland (Active Comparator): Each capsule contains 150 mg pregabalin.
  Interventions: Drug: Pregabalin capsules 150 mg of Pfizer Manufacturing Deutschland

INTERVENTIONS:
Drug: Pregabalin capsules 150 mg of Dexa Medica — Each capsule contains 150 mg of pregabalin. Test product was given as a single dose, under the procedure as described in the Section: Detailed description of the study.
  Other Names: Test product: pregabalin capsules 150 mg of Dexa Medica
  Arms: Pregabalin capsules 150 mg of Dexa Medica
Drug: Pregabalin capsules 150 mg of Pfizer Manufacturing Deutschland — Each capsule contains 150 mg of pregabalin. Reference product was given as a single dose, under the procedure as described in the Section: Detailed description of the study.
  Other Names: Reference product: Lyrica® 150 mg, produced by Pfizer Manufacturing Deutschland GmbH, Germany
  Arms: Pregabalin capsules 150 mg of Pfizer Manufacturing Deutschland

SUMMARY:
The present study was conducted to find out whether the bioavailability of 150 mg pregabalin capsules produced by Dexa Medica was equivalent to the reference products (Lyrica® capsule 150 mg, Pfizer Manufacturing Deutschland GmbH, Germany).

DETAILED DESCRIPTION:
This was a randomized, open label, two-period, two-sequence, crossover study under fasting condition. The participating subjects were required to have an overnight fast and in the next morning were given orally one capsule of the test drug (Pregabalin 150 mg produced by Dexa Medica) or one capsule of the reference drug (Lyrica® 150 mg, Pfizer Manufacturing Deutschland GmbH, Germany).

Blood samples were drawn immediately before taking the drug (control), at 20, 40 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24, 36 hours after drug administration. Seven days after the first drug administration (washout period), the procedure was repeated using the alternate drug. The plasma concentrations of pregabalin were determined by using validated liquid chromatography with tandem mass spectrometry detection (LC-MS/MS) method.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with absence of significant disease or clinically significant abnormal laboratory values or laboratory evaluation, medical history, or physical examination during the screening and could be considered healthy based on the evaluation
* Aged 18-55 years inclusive
* Preferably non-smokers or smoke less than 10 cigarettes per day
* Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study
* Body mass index within 18 to 25 kg/m2
* Vital signs (after 10 minutes rest) within the following ranges:

  * Systolic blood pressure: 100-120 mmHg
  * Diastolic blood pressure: 60-80 mmHg
  * Pulse rate: 60-90 bpm

Exclusion Criteria:

* Personal/family history of allergy or hypersensitivity or contraindication to pregabalin or allied drugs
* Pregnant or lactating women (urinary pregnancy test was applied to women subjects at screening and before taking the study drug)
* Any major illnesses in the past 90 days or clinically significant ongoing chronic medical illness e.g. congestive cardiac failure (heart failure), hepatitis, hypotensive episodes, hyperglycemia, etc
* Presence of any clinically significant abnormal values during screening, e.g. significant abnormality of liver function test (ALT, alkaline phosphatase, total bilirubin >= 1.5 ULN), renal function test (serum creatinine concentration > 1.4 mg/dL), etc
* Positive hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV
* Clinically significant electrocardiogram (ECG) abnormalities
* Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism, or excretion of the study drug, e.g. gastrointestinal disease including gastric or duodenal ulcers or history of gastric surgery
* Past history of anaphylaxis or angiodema
* History of drug or alcohol abuse within 12 months prior to screening for this study
* Participation in any clinical trial within the past 90 days calculated from the last visit
* History of any bleeding or coagulative disorders
* History of seizure, epilepsy, or any kind of neurological disorders
* History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm
* A donation or loss of 300 mL (or more) of blood within 3 months before this study's first dosing day
* Intake of any prescription, non-prescription drug, food supplements, or herbal medicines within 14 days of this study's first dosing day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUCt | 36 hours
  Area under plasma concentration time curve from time zero to the last observed quantifiable concentration was determined from plasma concentrations of pregabalin from the test drug and reference drug.
AUCinf | 36 hours
  Area under plasma concentration time curve from time zero to infinity was determined from plasma concentrations of pregabalin from the test drug and reference drug.
Cmax | 36 hours
  The peak plasma concentration of the drug was determined from plasma concentrations of pregabalin from the test drug and reference drug.
Tmax | 36 hours
  The time needed to achieve the peak plasma concentration was determined from plasma concentrations of pregabalin from the test drug and reference drug.

SECONDARY OUTCOMES:
T1/2 | 36 hours
  The elimination half life was determined from plasma concentrations of pregabalin from the test drug and reference drug.

CONTACTS AND LOCATIONS:
Overall Officials: Ratih SI Putri, MD, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia